CLINICAL TRIAL: NCT00115973
Title: An Open-Label, Stepwise Basal Insulin Dose Titration Study Using Continuous Subcutaneous Insulin Infusion (CSII) in Oral Antidiabetic Drug-Treated Type 2 Diabetes Mellitus Subjects Followed by a 10-Week Out-Patient Maintenance Phase
Brief Title: A Study of the Treatment of Type 2 Diabetes With an Insulin Infusion Pump
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDS253-1665
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Delivery Systems
Keywords: Pump; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: pump
Drug: insulin aspart

SUMMARY:
This trial is conducted in the United States of America (USA). This is an in-patient trial investigating stepwise dose increase in a period of up to 3-weeks followed by a 10-week out-patient maintenance period. A telephone contact visit is scheduled as a follow-up for the final clinic visit. A subject's participation in this trial would be expected to be up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosis at least 2 years ago
* Body Mass Index (BMI): 26-40 kg/m^2 (both inclusive)
* HbA1c: 7.5-10% (both inclusive)
* FPG values at least 140 mg/dl (7.8 mmol/l)

Exclusion Criteria:

* Use of drugs, which may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action or glucose utilization (steroids or non-specific beta-blockers)
* Current addiction to alcohol or substances of abuse or positive results on urine screen for drug and alcohol use
* Known or suspected allergy to trial products or related products

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-06; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 3 months

SECONDARY OUTCOMES:
Fasting plasma glucose
Plasma glucose profiles
Frequency of hypoglycemic events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (6):
- United States (6):
  - Novo Nordisk Investigational Site, Chula Vista, California
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Witchita, Kansas
  - Novo Nordisk Investigational Site, Willingboro, New Jersey
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, San Antonio, Texas

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com